CLINICAL TRIAL: NCT04771962
Title: Comparing the Efficacy Between Desflurane and Sevoflurane in Miantainance of Spontaneous General Anaesthesia Using Ambu Aura Gain in Paediatrics Patients
Brief Title: Comparison of the Anaesthetic Gases in Maintainance of General Anaesthesia in Paediatrics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Senior Consultant Anesthetist and lecturer, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USM/JEPem/18050248
Record Dates: First submitted 2020-11-04; First posted 2021-02-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Paediatrics; General Anaesthesia
Keywords: paediatrics; spontaneous general anaesthesia
MeSH Terms: interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DESFLURANE (Experimental): desflurane group- this group of patients will be induced with sevoflurane and maintained with desflurane during spontaneous general anaesthesia
  Interventions: Drug: DESFLURANE AND SEVOFLURANE
- SEVOFLURANE (Active Comparator): the controlled group.patients will be induced and maintained with sevoflurane through out spontaneous general anaesthesia.
  Interventions: Drug: DESFLURANE AND SEVOFLURANE

INTERVENTIONS:
Drug: DESFLURANE AND SEVOFLURANE — COMPARING THE EFFICACY IN MAINTAINANCE OF SPONTANEOUS GENERAL ANAESTHESIA USING AMBU AURA GAIN IN PEDIATRIC PATIENTS
  Other Names: Suprane and Sevoflurane

SUMMARY:
Desflurane and Sevoflurane are one of the modern inhalational anaesthetic agents currently in use in anaesthetic practice. The properties of desflurane that has low blood gas solubility coefficient of 0.47 compared to sevoflurane (0.68) made it more advantageous when used with supraglottic airway in maintaining general anaesthesia in paediatrics . It ensures rapid onset and offset of anaesthesia. Rapid recovery profiles especially among pediatric populations is to ensure less complications associated with prolonged recovery of anaesthesia upon emergence from anaesthesia. Nevertherless, desflurane has its drawback which is it can cause airway irritability related to its pungency. Hence, it is not used as an induction anaesthetic agent in paediatrics. This study was done to evaluate the effectiveness of desflurane in comparison to sevoflurane in maintaining spontaneous general anaesthesia in paediatrics population using Ambu AuraGain .

DETAILED DESCRIPTION:
Research design:

1. Double blinded , randomised controlled trial.
2. Involving paediatrics patients underwent elective surgeries requiring general anaesthesia in Hospital Universiti Sains Malaysia, Kubang Kerian.
3. The duration of the study is 24 months.

METHODOLOGY

1. After Approval from the Ethics Committee of University Sains Malaysia (USM), verbal and written consent will be taken from the patient's parent(s), 1 day prior of the surgery during pre-operative assessment in ward. All medical information of the patient will be kept confidential.
2. The study will be conducted to patient age 3 years to 12 years old, with body weight between 10-30kg after excluding patient who has a upper respiratory tract infection or known susceptible to malignant hyperthermia.
3. Patients who fulfil the inclusion and exclusion criteria during pre-operative assessment will be randomized into two group using computer generated randomization. The number generated will be placed in the envelope and allocation will be done on the day of the study prior to anaesthesia : S group (sevoflurane maintainance anaesthesia) = 40 and D group ( desflurane maintainance anaesthesia ) = 40.
4. Allocation concealment is being applied in this study to prevent selection bias by concealing the allocation sequence until the moment of assessing.
5. Participants and the researcher( whom assessing the outcomes ) are blinded during intervention ( double blinded ), where as the anesthetist in charge ( operator ) is not blinded.
6. Standard monitoring with non invasive blood pressure , electrocardiography capnography,and peripheral oxygen saturation ( SPO2) will be used.
7. Induction of anaesthesia with intravenous fentanyl 2mcg per kg, intravenous propofol of 2mg/kg and 3-4vol% of sevoflurane under 100% O2 mask ventilation.
8. The AmbuAuraGain will be used, with standard insertion technique.
9. After induction of anaesthesia, inhalation agent will be switch immediately according to group allocation for maintainance of anaesthesia.
10. Anaesthesia will be maintained using SEVOFLURANE at MAC of 1.2 to 1.5 for the S group and DESFLURANE at MAC 1.2 to 1.5 for the D group with mixture of oxygen/air mixture for both groups.
11. IV Paracetamol 15mg/kg and IV Fentanyl 0.5mcg/kg will be given as intraoperative analgesia.
12. Short acting opiod : IV fentanyl 0.5mcg per kg can be given as rescue analgesia.
13. At the end of surgery (the last suture put), the inhalational agents will be tapered down and discontinued, 100% oxygen with 6l/min was administered. The Ambu®AuraGain™ will be removed in the operating room once the child is fully awake (i.e: regular breathing, good tidal volume of 6-8ml/kg, gag reflex, grimacing and purposeful movements of the extremities).
14. The child then will be monitored in operating theatre recovery area until the modified Aldrete score reached 8.
15. Perioperative events in the operating room will be recorded by a blinded investigator. Any adverse events and emergence agitation during recovery will be recorded by a blinded nurse until patient is discharged to ward.
16. The first outcome of this study will be the intraoperative hemodynamics during maintainance of anaesthesia.
17. Baseline hemodynamic (blood pressure, heart rate, mean arterial pressure) of the patient during pre-intubation will be taken. After successful intubation, patient haemodynamics will be recorded at 10 minutes interval until 60 minutes and also during pre extubation and post extubation.
18. Second outcome will be the time of emergence ( the time interval from gas being off to patient awake,i.e: spontaneous eyes opening) , emergence agitation in recovery area, and the respiratory adverse events that occurs during maintainance of anaesthesia and emergence .
19. The respiratory events which will be recorded are, (ie: breath holding , bronchospasm, coughing, laryngospasm, copious secretions ( which required suctioning), desaturations ( SpO2 < than 90% ).

SAMPLE SIZE ESTIMATION

Objective 1 : hemodynamic changes ( heart rate)

To estimate the sample size for our study we utilized the G.Power sample size calculator software version 3.1 - Anova : repeated measures . Parametres used in the sample size are :

Effect size f : 0.39 ( for heart rate , Akhtam A. Shoukry et al,2016)

* 0.05 power : 0.80 number of groups: 2 number of measurements: 10 Standard Deviation within each group : 8.97 Mean group 1 : 68.04, mean group 2 : 75.09

Sample size is 32 per group. Estimated sample size with 10% drop out rate : 70

Objective 2 : Emergence time

To estimate the sample size for our study we utilized the PS: Power and Sample Size Calculations software,version 3.0. We applied the independent t-test. Parametres used in the sample size are :

Standard Deviation = 3.9 ( Demirbilek,2004) Mean difference = 3.8 ( expert opinion ) = 0.05 power = 0.80 m = 1 Sample size is 18 per group. Estimated sample size with 10% drop out rate :40

Objective 3 : Coughing on emergence

To estimate the sample size for our study, we utilized the PS: Power and Sample Size Calculations software,version 3.0. We applied the Dichotomous independent , two proportions,uncorrected chi-square test.

Parametres used in the sample size calculations are :

= 0.05, power = 0.80, m = 1, P0 = 0.49 ( proportion of desflurane among patients who did not cough), Paul at al,2010). P1 = 0.8 ( proportion of desflurane among patients who did cough,) expert opinion ).

Sample size is 36 per group.

Estimated sample size with 10% drop out rate : 80

STATISTICAL DATA ANALYSIS

OBJECTIVE 1:

numerical data will be analysed using ANOVA: repeated measures.

OBJECTIVE 2:

Numerical data will be analysed using independent t test.

OBJECTIVE 3:

Categorical data will be analysed using uncorrected chi square test.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 3 years to 12 years old.
* ASA (American Society of Anesthesiologist) I
* BMI (body mass index) less than 95 centile according to age, sex, height
* Preoperative assessment shows low risk of aspiration and no features of difficult intubation.
* No history of difficult intubation or history of admission to ICU for airway complication.
* Operation duration less or equal 2 hours using AmbuAuraGain.

Exclusion Criteria:

* Parent refusal for study participation to give informed consent.
* Patients who had an upper respiratory tract infection (URTI) within previous 2 weeks or any respiratory disease ( bronchial asthma, hyperactive airway,sleep apnea, chronic lung disease)
* Known susceptibility to malignant hyperthermia (MH)
* History of moderate to severe hepatic dysfunction following anaesthesia with desflurane not otherwise explained.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To compare the blood pressure intraoperatively between desflurane and sevoflurane. | up to 18 months
  by measuring the blood pressure
To compare the heart rate intraoperatively between desflurane and sevoflurane. | up to 18 months
  by measuring the heart rate
To compare the mean arterial pressure intraoperatively between desflurane and sevoflurane. | up to 18 months
  by measuring the mean arterial pressure

SECONDARY OUTCOMES:
To compare the emergence time ( interval from gas being off to patient awake). | up to 18 months
  to time how many minutes
To compare the respiratory events intraoperative and post operative | up to 18 months
  to observe for the signs :breath holding, bronchospasm,coughing, secretions,desaturations

CONTACTS AND LOCATIONS:
Overall Officials: Rhendra Hardy Mohamed Zaini, Principal Investigator — University Sains Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lerman J, Hammer GB, Verghese S, Ehlers M, Khalil SN, Betts E, Trillo R, Deutsch J; MAPS Investigators Group. Airway responses to desflurane during maintenance of anesthesia and recovery in children with laryngeal mask airways. Paediatr Anaesth. 2010 Jun;20(6):495-505. doi: 10.1111/j.1460-9592.2010.03305.x. Epub 2010 Apr 23. PMID 20456065
- [Background] Akhtam A. Shoukry, Ayman Abd Laltif,Amr Abd Fattah, Ibrahim Abd Ghani, Mohamed Serag. Isoflurane versus desflurane : hemodynamic parametres and recovery charecteristics:a comparative study.Ain Shams Journal of Anaesthesiology 2016,9:45-51
- [Background] Demirbilek S, Togal T, Cicek M, Aslan U, Sizanli E, Ersoy MO. Effects of fentanyl on the incidence of emergence agitation in children receiving desflurane or sevoflurane anaesthesia. Eur J Anaesthesiol. 2004 Jul;21(7):538-42. doi: 10.1017/s0265021504007069. PMID 15318465
- [Background] White PF, Tang J, Wender RH, Yumul R, Stokes OJ, Sloninsky A, Naruse R, Kariger R, Norel E, Mandel S, Webb T, Zaentz A. Desflurane versus sevoflurane for maintenance of outpatient anesthesia: the effect on early versus late recovery and perioperative coughing. Anesth Analg. 2009 Aug;109(2):387-93. doi: 10.1213/ane.0b013e3181adc21a. PMID 19608808
- [Background] Kim EH, Song IK, Lee JH, Kim HS, Kim HC, Yoon SH, Jang YE, Kim JT. Desflurane versus sevoflurane in pediatric anesthesia with a laryngeal mask airway: A randomized controlled trial. Medicine (Baltimore). 2017 Sep;96(35):e7977. doi: 10.1097/MD.0000000000007977. PMID 28858134
- [Background] Sethi S, Ghai B, Ram J, Wig J. Postoperative emergence delirium in pediatric patients undergoing cataract surgery--a comparison of desflurane and sevoflurane. Paediatr Anaesth. 2013 Dec;23(12):1131-7. doi: 10.1111/pan.12260. Epub 2013 Sep 19. PMID 24102666
- [Background] Davis PJ, Cohen IT, McGowan FX Jr, Latta K. Recovery characteristics of desflurane versus halothane for maintenance of anesthesia in pediatric ambulatory patients. Anesthesiology. 1994 Feb;80(2):298-302. doi: 10.1097/00000542-199402000-00009. PMID 8311312
- [Background] Jindal R, Kumra VP, Narani KK, Sood J. Comparison of maintenance and emergence characteristics after desflurane or sevoflurane in outpatient anaesthesia. Indian J Anaesth. 2011 Jan;55(1):36-42. doi: 10.4103/0019-5049.76604. PMID 21431051
- [Background] Satyanarayana A, Aparanji K, Gopalakrishna K. Comparison of airway responses, haemodynamics and recovery using sevoflurane and desflurane via laryngeal mask airway in day care paediatric surgeries. J. Evid. Based Med. Healthc. 2017; 4(92), 5559-5563.
- [Background] Kotwani MB, Malde AD. Comparison of maintenance, emergence and recovery characteristics of sevoflurane and desflurane in pediatric ambulatory surgery. J Anaesthesiol Clin Pharmacol. 2017 Oct-Dec;33(4):503-508. doi: 10.4103/joacp.JOACP_194_16. PMID 29416244